CLINICAL TRIAL: NCT03746938
Title: First Open-label Trial in Humans to Evaluate the Safety and Efficacy of Epicardial Delivery of Collagen Patches With Adipose-derived Stem Cells in Patients With Ischemic Heart Disease and Left Ventricular Dysfunction.
Brief Title: First in Humans to Evaluate Collagen Patches With Stem Cells in Patients With Ischemic Left Ventricular Dysfunction
Acronym: CARDIOMESH
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Viscofan (Industry)
Collaborators: Ministerio de Ciencia e Innovación, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARDIOMESH
Record Dates: First submitted 2018-11-13; First posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Heart Failure With Reduced Ejection Fraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VB-C01 (Experimental): Surgical technique: Via left lateral thoracotomy, the heart is lifted and supported on two deep pericardial points with 4-0 or 5-0 Prolene double arrmed suture. Each suture is passed through the reinforced frame of the collagen membrane containing the stem cells (VB-C01) and then tied, while the upper part of the patch is held with forceps. After securing the lower part of the pericardial layer, the heart is allowed to slowly recover its position with the pericardial cavity while the collagen membrane is mobilized to cover all of the target area. If necessary, some sutures can be used to fix the patch VB-C01 to the epicardial surface of the heart. Each suture is likewise passed through the reinforced frame of the membrane.
  Interventions: Device: VB-C01

INTERVENTIONS:
Device: VB-C01 — Surgical implant of VB-C01 (Collagen membrane seeded with allogeneic stem cells isolated from adipose tissue, ADSC).

SUMMARY:
It´s a first open-label trial in humans to evaluate the safety and efficacy of epicardial delivery of collagen patches with adipose-derived stem cells in patients with ischemic heart disease and left ventricular dysfunction that remain symptomatic despite optimal medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥18 years and ≤80 years.
* LVEF ≤35% as assessed by echocardiography, confirmed by MRI if there are no contraindications for this procedure.
* History of revascularised or nonrevascularisable coronary artery disease as the cause of ventricular dysfunction.
* NYHA functional class III for dyspnea under optimal medical treatment.
* Ability to perform the exercise test with respiratory gas consumption. MVO2 should be ≥ 10 and ≤ 18 ml/kg/min in the exercise test.
* Ability to perform a 6-minute walk test > 100 m and ≤ 400 m.
* Haemodynamic stability (blood pressure > 100/40 mmHg, heart rate < 110 bpm and oxygen saturation at rest in room air > 95%).

Exclusion Criteria:

* Participation in another clinical trial within 30 days prior to inclusion.
* Prior treatment with cell or gene therapy.
* Diagnosis of acute myocardial infarction with 3 months prior to inclusion.
* Significant coronary artery disease eligible for revascularization.
* Significant valvular disease eligible for surgery.
* Presence of uncontrolled ventricular arrhythmias (VR or VF) at the time of implant surgery.
* Women who are pregnant or breastfeeding.
* Mental disease or psychological condition that impedes the subject from understanding the nature of the protocol and granting his/her consent.
* Advanced dementia according to the Barthel index.
* Active systemic infection.
* History of primary or acquired immunodeficiency or on immunosuppressive therapy (within 3 months prior to inclusion or if the need for immunotherapy is foreseeable at any time during the study follow-up).
* Tumour disease, except that eradicated at least 5 years prior to inclusion in the study and without receiving chest radiotherapy. Completely eradicated nonmelanoma skin tumours (at any time) not requiring chest chemotherapy or radiotherapy) are permitted.
* History of autoimmune disease.
* Stroke within 12 months prior to inclusion.
* Respiratory compromise or need for home oxygen therapy.
* Life expectancy of less than 1 year for any reason.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-11-13 (Estimated); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Composite safety endpoint formed by the major adverse cardiac and cerebrovascular events (MACCE) occurring on all visits during the first year after implantation. | During the first year after implantation
  MACCE include: all-cause death, cardiovascular death, re-infarction, need for revascularization, hospitalization for heart failure, sustained ventricular tachycardia, ventricular fibrillation, or stroke.

SECONDARY OUTCOMES:
Incidence of all-cause death | During the first year after implantation
Incidence of cardiovascular death | During the first year after implantation
Incidence of re-infarction | During the first year after implantation
Incidence of need for revascularization | During the first year after implantation
Incidence of hospitalization for heart failure | During the first year after implantation
Incidence of sustained ventricular tachycardia | During the first year after implantation
Incidence of ventricular fibrillation | During the first year after implantation
Incidence of stroke | During the first year after implantation
Incidence of surgical complications | During the first year after implantation
Changes in the pericardial physiology | During the first year after implantation
  Assessed by echocardiography or MRI
VT inducibility | During the first year after implantation
  Heterogeneous tissue on MRI as well as the presence of late potentials on the electrophysiological study scheduled at 1 year of follow-up.
Changes in DSA-HLA | During the first year after implantation
Changes in proinflammatory cytokines | During the first year after implantation
Changes in immunological cell types. | During the first year after implantation
Changes in end-systolic volume | During the first year after implantation
  Measured by echocardiography comparing the baseline study of each patient with the studies performed in that same patient during the follow-up.
Changes in end-diastolic volume | During the first year after implantation
  Measured by echocardiography comparing the baseline study of each patient with the studies performed in that same patient during the follow-up.
Changes in left ventricular ejection fraction | During the first year after implantation
  Measured by echocardiography comparing the baseline study of each patient with the studies performed in that same patient during the follow-up.
Changes in sphericity index | During the first year after implantation
  Measured by echocardiography comparing the baseline study of each patient with the studies performed in that same patient during the follow-up.
Changes in segmental contraction score (normal / hypokinetic / akinetic / dyskinetic) in the 17 myocardial segments | During the first year after implantation
  Measured by echocardiography comparing the baseline study of each patient with the studies performed in that same patient during the follow-up.
Changes in systolic thickening by myocardial segments | During the first year after implantation
  Measured by echocardiography comparing the baseline study of each patient with the studies performed in that same patient during the follow-up.
Changes in the scar size expressed in grams | During the first year after implantation
  Measured by MRI comparing the baseline study of each patient with the studies performed in that same patient during the follow-up.
Changes in the viable myocardial mass expressed in grams | During the first year after implantation
  Measured by MRI comparing the baseline study of each patient with the studies performed in that same patient during the follow-up.
Changes in the scar size expressed in percentage of LV | During the first year after implantation
  Measured by MRI comparing the baseline study of each patient with the studies performed in that same patient during the follow-up.
Changes in the percentage of viable myocardium in LV | During the first year after implantation
  Measured by MRI comparing the baseline study of each patient with the studies performed in that same patient during the follow-up.
Changes in the functional class | During the first year after implantation
  According to the New York Heart Association (NYHA) for dyspnea
Changes in the patient-perceived quality of life | During the first year after implantation
  According to the Minnesota Living with Heart Failure Questionnaire (MLHFQ)
Changes in the distance covered on the 6-minute walk test | During the first year after implantation
Changes in the peak oxygen consumption on ergospirometry | During the first year after implantation
Changes in the brain natriuretic peptide | During the first year after implantation

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Jesús Fernández-Avilés Díaz, Principal Investigator — Hospital General Universitario Gregorio Marañón
Locations (2):
- Spain (2):
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital General Universitario Gregorio Marañón, Madrid

IPD SHARING:
Plan to Share IPD: Undecided